CLINICAL TRIAL: NCT01185834
Title: Assessment of Lotrafilcon A Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: P-335-C-015
Record Dates: First submitted 2010-08-18; First posted 2010-08-20 (Estimated); Results first posted 2012-01-24 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2011-12

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Device: Lotrafilcon A upgrade soft contact lens — Silicone hydrogel contact lens approved for daily wear and extended wear up to 30 consecutive nights.

SUMMARY:
The purpose of this 3-month study is to evaluate subjective responses to an upgraded contact lens.

ELIGIBILITY:
Inclusion Criteria:

* Have normal ocular findings.
* Be able to wear the study lenses in the available powers.
* Currently wear contact lenses for a minimum of 5 days a week, and at least 8 hours a day.
* Wear Night & Day contact lenses.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Require concurrent ocular medication.
* Eye injury or surgery within twelve weeks prior to enrollment.
* Currently enrolled in an ophthalmic clinical trial.
* Any active corneal infection.
* Corneal refractive surgery.
* Wear AIR OPTIX NIGHT & DAY AQUA lenses.
* Other protocol-defined exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2010-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirteen US optometry sites recruited and enrolled subjects for this study.
Groups:
- Lotrafilcon A: Lotrafilcon A lenses worn for 3 months, replaced monthly. Lenses worn on the same basis as habitual lenses, as prescribed by eye care practitioner (e.g., daily wear, flexible wear, extended wear up to 30 continuous nights).
Period: Overall Study
Arm/Group | Lotrafilcon A
Started | 118
Completed | 104
Not Completed | 14
Not completed — Lost to Follow-up | 2
Not completed — Discomfort | 4
Not completed — Biomicroscopy | 4
Not completed — Time/Job Conflict | 2
Not completed — Early exit - Site error | 2

BASELINE CHARACTERISTICS:
Arm/Group | Lotrafilcon A
Number analyzed (Participants) | 118
Age Continuous [Mean (Standard Deviation); unit: years] | 34.1 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84
  Male | 34

OUTCOME MEASURES:

1. Primary Outcome: Overall Comfort
Description: As interpreted by the participant and recorded on a questionnaire as a single, retrospective evaluation of 3 months of wear time. Overall comfort was evaluated binocularly and rated on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 3 months of wear, replacing lenses monthly
Population: Analysis conducted per protocol, with exclusions due to reasons such as: major protocol deviations as determined by masked review; discontinuations; and/or missing responses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lotrafilcon A
Number analyzed (Participants) | 103
units on a scale | 8.4 (1.6)

2. Secondary Outcome: Overall Lens Fit
Description: As assessed by the investigator at study visit using a biomicroscope, which magnifies the appearance of the contact lens on the participant's eye. Lens fit was graded by eye on a 5-point scale, with 2=unacceptably loose, 1=acceptably loose, 0=optimal, -1=acceptably tight, and -2=unacceptably tight
Time Frame: 3 months of wear, replacing lenses monthly
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Lotrafilcon A
Number analyzed (Participants) | 103
Number analyzed (Eyes) | 206
units on a scale | 0.0 (0.3)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of the trial: 143 days.
Description: This reporting group includes all enrolled and exposed participants.
Arm/Group | Lotrafilcon A
Serious Adverse Events (participants affected / at risk) | 0/118
Other Adverse Events (participants affected / at risk) | 0/118

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.